CLINICAL TRIAL: NCT04148703
Title: Cost-utility Analysis of the Follow-up of Exclusive Telemedicine Pacemakers, Compared to Conventional Pacemakers
Acronym: TELEPACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Tours University Hospital (Unknown); University Hospital, Marseille (Other); Rennes University Hospital (Other); University Hospital, Toulouse (Other); University Hospital, Clermont-Ferrand (Other); Angers University Hospital (Unknown); Lille University Hospital (Unknown); University Hospital, Strasbourg, France (Other); University Hospital, Rouen (Other); Montpellier University Hospital (Unknown); University Hospital, Brest (Other); Pau University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC18_0431
Record Dates: First submitted 2019-10-24; First posted 2019-11-01 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Single or Dual Chamber Pacemaker Implantation; Home Monitoring Follow-up
Keywords: Pacemaker, home monitoring, remote monitoring, ecocomic
MeSH Terms: interventions — Working Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Experimental): in-office follow-up at 30 days post-implantation and after by remote monitoring (daily) without scheduled in-office follow-up during the study period (48 months). A remote FU will be planned every 9 months.
  Interventions: Other: Follow up post Pacemaker implantation by home monitoring
- Control group (Active Comparator): The patients randomized in the control group will be followed accordingto the guidelines; i.e. with an in-office follow-up at 30 days post-implantation and after followed with in-office follow-ups according to clinical practice.
  Interventions: Other: Follow up post Pacemaker implantation in office

INTERVENTIONS:
Other: Follow up post Pacemaker implantation in office — All patients will be implanted with a single or dual chamber pacemaker according the implantation guidelines and will be followed by in-office follow-up
  Arms: Control group
Other: Follow up post Pacemaker implantation by home monitoring — All patients will be implanted with a single or dual chamber pacemaker according the implantation guidelines and will be followed by home monitoring
  Arms: Active group

SUMMARY:
TELEPACE is an economic evaluation that aims to determine the probability at which Home Monitoring without physical examinations, could be cost effective, compared to the conventional treatment by face to face consultations. Patient will be randomized in a control group followed according to the current guidelines and and active group exclusively followed by remote monitoring. The study will end after a 4 year follow-up.

DETAILED DESCRIPTION:
Professional practice guidelines recommend that pacemakers be followed with at least one to two in-office follow-ups per year, which is both a public health issue (the average time to get a consultation with a cardiologist being 42 days) but also an economic issue considering the number of patients implanted (Brignole EHJ 2013). Remote monitoring of pacemakers could allow an optimization of the long-term follow-up of pacemaker recipients in hospitals.

Compared to CRT and ICD, few studies have highlighted the economic advantage of remote monitoring with PM.

COMPAS study (Eur Heart J. 2012) demonstrated that remote monitoring is a safe alternative to conventional care over a 2 year-follow-up. This study also demonstrated that long-term remote monitoring of pacemakers decreased the number of ambulatory visits and enabled the early detection of important clinical and device-related adverse events.

As the study shows data up to 18 months, this is not sufficient to define the benefit of telecardiology in this population of patients.

SETAM study (Pacing Clin Electrophysiol 2017) demonstrated the benefit of remote monitoring showing an earlier diagnosis and management of atrial arrhythmias and a subsequently reduction of atrial fibrillation (AF) burden. The incidence and prevalence of AF is expected to increase with time, resulting in significant societal and economic impact.

Neither COMPAS nor SETAM were designed as economic evaluations

TELEPACE study proposes the first economic evaluation of an exclusive follow-up by Home-Monitoring of patients implanted with pacemaker for a period of 4 years.

All patients will be implanted with a single or dual chamber pacemaker according the implantation guidelines. Patients enrolled will be then randomized to a control group or an active group:

* The patients randomized in the control group will be followed accordingto the guidelines; i.e. with an in-office follow-up at 30 days post-implantation and after followed with in-office follow-ups according toclinical practice.
* Active group: in-office follow-up at 30 days post-implantation and after by remote monitoring (daily) without scheduled in-office follow-up during the study period (48 months). A remote FU will be planned every 9 months.

Consequently, compared to the guidelines, the patients in the active group will be followed according to the guidelines; except for the in-office follow-ups annually.

By collecting real costs directly on health insurance reimbursement bases (SNIIRAM), this study will define the medico-economic benefit of remote monitoring of pacemakers.

A cost-utility analysis is needed to address the question. The use of QALYs is not intended to demonstrate a difference in clinical efficacy but to ensure that efficacy and costs are studied simultaneously which is required in order to avoid risk inflation when differences in efficacy and costs are studied sequentially.

If there is no significant differences in QALYs (as expected) but there are savings in terms of HSR then the cost-utility ratio will allow to estimate a "net benefit criterion" (NBC) that translates QALYs into money as follows: NBC = WTP.(differences in QALYs) - (differences in costs) where WTP represents the (societal) willingness to pay a QALY.

If there is no differences in QALYs the NBC will then reduce to a cost-minimisation calculus (WTP.(diff QALYs) = 0).

Cost-minimisation alone can only be used (HAS regards it as a sub-category of cost-effectiveness analysis whose use has to be duly justified) provided that there is strong evidence of equivalence in terms of clinical efficacy. If this is not the case, a cost-utility analysis will be more relevant as it will test simultaneously for both differences in efficacy and in costs.

Moreover, the study will confrim the safety of telecardiology and evaluate patients' individual preferences for the different management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Single or dual chamber pacemaker implantation patients
* patients agree to be enrolled in the study and followed during 4 years
* patients have insurance coverage

Exclusion Criteria:

* Minor patients
* personn with disability
* pregnant women
* patient with life expectancy of less than 4 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
ICER (incremental cost effectivness ratio) | 4 years
  cost and medical consumtion collected with the French insurance care database
QALY | 4 years
  Quality Adjusted Life Years estimated by EQ5D-5L

SECONDARY OUTCOMES:
Safety of home monitoring | 4 years
  time limit compensation claim (delay between the diagnosis and the therapy)
Safety of home monitoring | 4 years
  combined criteria (death, stroke, heart failure, arrhythmia, pacemeker dysfunction, infection, hospitalization)

CONTACTS AND LOCATIONS:
Locations (1):
- GOURAUD Jean-Baptiste, Nantes, France